CLINICAL TRIAL: NCT06002412
Title: Deep Learning-based Quality Control of Ultrasound Images During Early Pregnancy
Brief Title: Quality Control of Ultrasound Images During Early Pregnancy Via AI
Status: Recruiting | Type: Observational
Sponsor: Chinese Academy of Sciences (Other Government)
Collaborators: Beijing Obstetrics and Gynecology Hospital (Other); Peking University Third Hospital (Other); Changsha Hospital for Maternal and Child Health Care (Other); Second Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Di Dong, Professor, Chinese Academy of Sciences
Other Study IDs: CASMI005
Record Dates: First submitted 2023-08-13; First posted 2023-08-21 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Early Pregnancy
Keywords: Early Pregnancy; Ultrasound; Quality Control

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Beijing Obstetrics and Gynecology Hospital affiliated to Capital Medical University: Beijing Obstetrics and Gynecology Hospital affiliated to Capital Medical University collects clinical information and ultrasound images of sagittal, NT and choroid plexus views of the fetus which was obtained from early pregnant women who underwent NT sweeps.
  Interventions: Other: Image quality control
- Peking University Third Hospital: Peking University Third Hospital collects clinical information and ultrasound images of sagittal, NT and choroid plexus views of the fetus which was obtained from early pregnant women who underwent NT sweeps.
  Interventions: Other: Image quality control
- Changsha Hospital for Maternal and Child Health Care: Changsha Hospital for Maternal and Child Health Care collects clinical information and ultrasound images of sagittal, NT and choroid plexus views of the fetus which was obtained from early pregnant women who underwent NT sweeps.
  Interventions: Other: Image quality control
- Second Xiangya Hospital of Central South University: Second Xiangya Hospital of Central South University collects clinical information and ultrasound images of sagittal, NT and choroid plexus views of the fetus which was obtained from early pregnant women who underwent NT sweeps.
  Interventions: Other: Image quality control

INTERVENTIONS:
Other: Image quality control — The investigators identify the region of interest in the relevant section to give a conclusion on whether the image is standard or not, guiding clinicians to standardize the operation, and reducing the rate of misdiagnosis and underdiagnosis.

SUMMARY:
This research integrates artificial intelligence to enhance early pregnancy ultrasonography quality control, focusing on specific fetal sections. In collaboration with prominent medical institutions, the investigators have amassed extensive fetal ultrasound data. The investigators aim to develop a deep learning model that can accurately identify essential anatomical areas in ultrasound images and evaluate their quality. This tool is expected to significantly decrease misdiagnoses of conditions like Down Syndrome and neural system deformities by ensuring real-time image quality assessment.

DETAILED DESCRIPTION:
This research is dedicated to integrating artificial intelligence technology to optimize the quality control process of early pregnancy ultrasonography. The ultrasound images involved primarily focus on the median sagittal section, NT section, and choroid plexus of the fetus during early pregnancy. In this regard, the investigators have collaborated with renowned medical institutions such as Beijing Obstetrics and Gynecology Hospital, Peking University Third Hospital, Changsha Hospital for Maternal and Child Health Care, and Second Xiangya Hospital of Central South University to retrospectively and prospectively collect a vast amount of early pregnancy fetal ultrasound image data. Based on this, the investigators plan to establish a model rooted in deep learning. This model will be capable of precisely identifying key anatomical regions in standard ultrasound scan images. Furthermore, by recognizing these anatomical structures, the model will determine whether the ultrasound image meets the standard scanning quality. This model is anticipated to serve as a powerful auxiliary tool in obstetric ultrasonography, enabling real-time assessment of ultrasound image quality, thereby significantly reducing the rates of missed and misdiagnosed fetal diseases such as Down Syndrome and neural system malformations.

ELIGIBILITY:
Inclusion Criteria:

* Women in early pregnancy who have detailed personal information and ultrasound images.
* The ultrasound images should clearly show the fetus's median sagittal, NT, and choroid plexus views.

Exclusion Criteria:

* Ultrasound images from women in mid to late pregnancy.
* Ultrasound images that are unclear or blurry, making evaluation difficult.
* Women who did not provide complete personal and medical information during the ultrasound scan.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women in early pregnancy
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2028-07-30 (Estimated)

PRIMARY OUTCOMES:
PR curve of image quality control module | one month
  Using Precision-Recall curve and mean average percision as evaluating indicator of image quality control model.

SECONDARY OUTCOMES:
The accuracy of intelligent analysis system in image quality control module | one month
  The agreement between the prediction outcome of intelligent analysis system and the golden standard

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Beijing Obstetrics and Gynecology Hospital affiliated to Capital Medical University, Beijing
  - Peking University Third Hospital, Beijing
  - Changsha Hospital for Maternal and Child Health Care, Changsha
  - Second Xiangya Hospital of Central South University, Changsha

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) may be made available to other researchers upon request. Interested researchers should present a reasonable research proposal and a data usage application. All participating units of this study will review and assess the proposal and application to determine whether to share the data.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will become available 6 months after study completion and will remain available for a period of 5 years.
Access Criteria: Interested researchers should submit a detailed research proposal and a data usage application for review. All participating units of this study will assess the application to determine eligibility for data access.
URL: http://www.radiomics.net.cn/